CLINICAL TRIAL: NCT00953225
Title: Vitamin D Supplementation in Veterans With Early-Stage Prostate Cancer
Acronym: vit D & PCa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-004-09S; MUSC IRB HR#19344 (Other: MUSC IRB)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; vitamin D
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D3 (Experimental): 4,000 IU vitamin D3 daily for one year
  Interventions: Drug: vitamin D3
- Placebo (Placebo Comparator): Placebo daily for one year
  Interventions: Drug: Placebo daily for one year

INTERVENTIONS:
Drug: vitamin D3 — 4,000 IU daily for one year
  Arms: Vitamin D3
Drug: Placebo daily for one year — Placebo
  Arms: Placebo

SUMMARY:
Vitamin D promotes the differentiation of prostate cancer cells, maintains the differentiated phenotype of prostate epithelial cells, and can induce prostate cancer cell death, raising the possibility that vitamin D deficiency over time promotes the progression of subclinical prostate cancer to clinical disease. The investigators propose to conduct a clinical study aimed at measuring the efficacy of vitamin D3 (4000IU/day) supplementation in Veterans diagnosed with low-risk, early-stage prostate cancer, who elect to have their disease monitored through active surveillance. The successful completion of this proposed clinical study will allow us to determine whether correcting vitamin D deficiency in Veterans diagnosed with early-stage prostate cancer will prevent progression of their disease and improve their prognosis.

DETAILED DESCRIPTION:
Vitamin D promotes the differentiation of prostate cancer (PCa) cells, maintains the differentiated phenotype of prostate epithelial cells, and can induce prostate cancer cell death, raising the possibility that vitamin D deficiency over time promotes the progression of subclinical PCa to clinical disease. These considerations support the use of vitamin D3 as a chemopreventive agent.

We hypothesize that a daily dose of vitamin D3 (4,000 IU) taken for one year by Veterans diagnosed with low-risk, early-stage PCa, who are eligible for active surveillance will: a) result in a measurable decrease of serum PSA levels in a significant number of enrolled subjects, and b) be associated with a stabilization or improvement of their PCa pathology, as assessed through histological examination of prostate tissue biopsy specimens (Gleason score and percent of positive biopsies) obtained at the end of the study, as part of their standard medical care for active surveillance.

This VA Merit application proposes to conduct a randomized, placebo-controlled clinical study aimed at measuring the efficacy of vitamin D3 (4000IU/day) supplementation in Veterans diagnosed with early-stage prostate cancer, who elect to have their disease monitored through active surveillance (before considering definitive therapy). The main objectives of this proposed clinical study are as follows:

1. To determine whether a daily supplement of 4,000 IU of vitamin D3 taken for twelve months will result in a measurable and significant decrease of serum PSA levels in Veterans diagnosed with low-risk, early stage PCa (Gleason score 6, PSA 10, clinical stage T1C or T2a), who elect to have their disease monitored through active surveillance for at least one year.
2. To determine in enrolled Veterans the pathology status of their PCa by analyzing prostate tissue biopsy specimens at the end of the study (Gleason score and percentage of positive biopsies), and by comparing them with those obtained before enrollment in this study, as part of their standard medical care.

The implementation of these proposed studies will allow us to assess whether vitamin D3 supplementation can be utilized as a chemopreventive regimen in Veterans diagnosed with low-risk, early stage PCa, and provide a useful addition to active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Male Veterans (> 18 years of age) recently diagnosed with low-risk PCa (histologically documented adenocarcinoma of the prostate)
* A serum PSA value of up to 10.0 ng/ml, and a Gleason score of six or less (three or less in either architectural pattern)
* For the purpose of eligibility, these additional criteria will be verified: *serum creatinine 2.0 mg/dL

  * serum phosphate (measured as phosphorus) > 2.3 and < 4.8 mg/dL
  * serum calcium > 8.5 and < 10.5 mg/dL

Exclusion Criteria:

* Subjects with any concurrent malignancy, except non-melanoma skin cancer
* Subjects with a history of sarcoidosis
* Subjects with a history of high-dose (1,000 IU per day) vitamin D supplementation
* Subjects with a history of hypercalcemia
* Subjects who use lithium as a medication

Ages: 19 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — diagnosis of early-stage prostate cancer
Enrollment: 83 (Actual)
Dates: Start 2010-01-07 (Actual); Primary Completion 2013-12-15 (Actual); Study Completion 2014-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Gattoni-Celli, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (2):
- United States (2):
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was based in the Urology Clinics at the Medical University of South Carolina (MUSC) and the Charleston VA Medical Center, and the MUSC Radiation Oncology Clinic, all located in Charleston, SC. The recruitment period was from October 2010 through December 2012.
Period: Overall Study
Arm/Group | Vitamin D3 | Placebo
Started | 46 | 37
Completed | 44 | 37
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 | Placebo | Total
Number analyzed (Participants) | 46 | 37 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 19 | 44
  >=65 years | 21 | 18 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 46 | 37 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 46 | 37 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 18 | 36
  White | 27 | 19 | 46
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PSA Slope (Trajectory) or the Change in PSA Level Over Time
Description: Change in PSA (ng/mL) from baseline to 1 year visit, which include the baseline through 1 year follow-up.
Time Frame: 1 year (visits # 1-8)
Population: Linear regression was applied to each subject's data with Log(PSA +1) as the outcome. Based on the fitted model, the change in PSA from visit #1 (baseline) to visit #8 (1 year) was calculated. This derived change score is summarized by group.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 44 | 37
ng/mL | 0.59 [-0.20 to 1.44] | 0.27 [-0.57 to 1.64]

2. Secondary Outcome: Number of Positive Biopsy Cores (Out of Twelve) Compared to the Corresponding Values Assessed Before Enrollment
Description: Change in the number of positive cores per subject from the pre-study prostate biopsy to the repeat prostate biopsy following study participation.
Time Frame: 1 year
Population: Each subject had 12 cores measured at each of the pre and post prostate biopsies. The variable summarized is the number of positive cores per subject.
Measure: Median (Inter-Quartile Range); unit: cores per subject
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 42 | 35
cores per subject | -1.00 [-1.00 to 0.25] | 0.00 [-1.00 to 1.00]

ADVERSE EVENTS:
Time Frame: The Recruitement Period was OCT 2010 - DEC 2012. Final particpant study visit was OCT 2013. Adverse Event data was collected over a period of 3 years.
Groups:
- Arm 1: 4,000 IU vitamin D3 daily for one year
  vitamin D3: 4,000 IU daily for one year
- Arm 2: Placebo daily for one year
  Placebo daily for one year: Placebo
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/37
Other Adverse Events (participants affected / at risk) | 0/46 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No